CLINICAL TRIAL: NCT02263820
Title: Novel Biomarkers for Risk Prediction of Contrast-Induced Acute Kidney Injury Post Coronary Angiography (NORDICA Study)
Brief Title: Novel Biomarkers for Risk Prediction of Contrast-Induced Acute Kidney Injury Post Coronary Angiography
Acronym: NORDICA
Status: Completed | Type: Observational
Sponsor: Sapere Bio (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: HSDX-1502
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Acute Kidney Injury; Renal Insufficiency; Kidney Diseases
Keywords: Acute Kidney Injury; Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, plasma, buffy coat
Oversight: Data Monitoring Committee: No

SUMMARY:
Contrast-induced acute kidney injury (CI-AKI) has been recognized as the third most common cause of hospital acquired AKI, after hypotension-associated hypo-perfusion and post-operative AKI. The development of CI-AKI after cardiac catheterization is associated with a significant increase in both short-term and long-term mortality and morbidities, as well as an increase in length of stay and cost.

The only marker of renal function that has predictive ability is creatinine and it has significant limitations in identifying patients who will develop AKI. Therefore, a diagnostic test for predicting CI-AKI risk would have widespread clinical utility.

The primary purpose of this study is to measure the association between baseline expression of senescence markers in blood using SenesceTest and the occurrence of CI-AKI post cardiac catheterization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 yo) undergoing invasive coronary angiography with or without percutaneous coronary intervention (PCI), that are predicted to have ≥14% risk of developing AKI as defined by Mehran et al.
* Medically compliant and able to consent and follow detailed directions
* Agree to additional collection of blood sample 48-72h post cardiac catheterization

Exclusion Criteria:

* Presence of acute, active infection (e.g. HIV, pneumonia, septic shock).
* Contrast media exposure within last 48h
* Presenting with systolic time-segment elevation myocardial infarction.
* Presence of cardiogenic shock
* Presence of hemodynamic instability or requiring pressors or intra-aortic balloon pump
* Severe kidney disease with estimated glomerular filtration rate <30 mL/min/1.73m2 or receiving dialysis for end stage renal disease
* Kidney transplant and liver transplant patients and all patients currently on immunosuppressants
* Severe heart failure with known ejection fraction <25%
* Prior heart transplant
* Chronic liver disease /cirrhosis
* Patients actively undergoing chemotherapy or radiation treatment for any indication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing cardiac catheterization with or without percutaneous coronary intervention (PCI)
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in serum creatinine levels (absolute and percentage) | Measured 48-72h after catheterization

SECONDARY OUTCOMES:
Major Adverse Clinical Events (MACE, a composite of all-cause mortality, myocardial infarction or renal replacement therapy) | Within 90 days after catheterization
Admission to the ICU | Within 90 days after catheterization

CONTACTS AND LOCATIONS:
Overall Officials: George A Stouffer, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Heart & Vascular Care, Chapel Hill, North Carolina, United States